CLINICAL TRIAL: NCT03511742
Title: Functional Characteristics of ICUs in Uganda and Their 28-day Patient Mortality
Brief Title: Functional ICUS in Uganda and Their Survival Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Resident Anesthesia and critical care, Makerere University
Other Study IDs: #REC REF 2018-004
Record Dates: First submitted 2018-04-10; First posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study is to describe the functional characteristics of Icus in Uganda and their @8-day patient characteristics it is a prospective cohort study .All Icus in Uganda will be included and their admitted patients followed upto 28 days in the ICU for mortality

DETAILED DESCRIPTION:
Intensive Care units are specialized units with expertise to provide organ support for the critically ill patients. There's a growing global burden of critical illness especially in the low-income coun-tries where critical care services are limited. Despite advances in critical care, the mortality in Uganda remains very high, with sepsis and trauma as the major contributors. There's paucity of literature regarding ICUs characteristics, disease burden and patient characteristics which could be contributing to the high mortality.

Objectives To describe the functional characteristics of the ICUs in Uganda. To determine the ICU mortality of critically ill patients in Uganda. To determine the risk factors of mortality of patients admitted in the ICU Methods A prospective cohort study will be carried out in all ICUs in Uganda. All new patients in the ICUs will be recruited into the study. Data will be collected onto two separate questionnaires, one for patient characteristics and the second for ICU functional characteristics. The patient's data will be collected within the first 24 hours and patients will be followed up for death\discharge within 28 days in the ICU. The data will be collected from the patients' charts and entered into Epidata.

ELIGIBILITY:
Inclusion Criteria:

All new patients admitted to Uganda's Intensive Care Units ICUs in Uganda whose unit heads verbally consent to participate in the study.

Exclusion Criteria:

Patients transferred in from another unit will not be re recruited. ICUs that don't consent to the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Target population Critically ill patients in all Intensive care units in Uganda Accessible population. All ICUs in Uganda. All patients admitted to the intensive care units in Uganda during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
28 day mortality | 3 months
  Total number of patients who died during the study period within 28 days over the total number recruited, and a survival analysis will be plowed on a Kaplan Meier
functional characteristics of ICUs in Uganda | 3 months
  outcome measure will be descriptive, that is interms of ICU location(urban or rural), staffing (nurse to patient ratio), infrastructure(floor space cm2), monitoring equipment, services rendered(organ support), and the ICU operation models(closed versus open) will be assessed for association with patient outcome

SECONDARY OUTCOMES:
factors associated with mortality | 3 months
  Age ( years), sex, indication for admission, length of ICU stay(days), comorbidities, HIV and HAART status, Mechanical ventilation(days) and length on ICU stay(days), ICU final diagnosis, Ino-tropic/vasopressor use, Sedation, NEWS score will be run in univariate and multivariate to assess association with mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Atumanya Patience, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
analyses data will be published in a peer reviewed journal
Supporting Information: SAP, CSR, Analytic Code
Time Frame: within 6 months
Access Criteria: open access